CLINICAL TRIAL: NCT04777227
Title: Effectiveness of Saline Water and Lidocaine Injections for the Treatment of Intractable Plantar Keratoma: A Randomised Feasibility Study
Brief Title: Effectiveness of Saline Water and Lidocaine Injections for the Treatment of Intractable Plantar Keratoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Vincent Cantin, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Intractable Plantar Keratoma
MeSH Terms: interventions — Lidocaine; Debridement

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Debridement (Active Comparator): A debridement (procedure involving cleaning and removing all hyperkeratotic tissue) was completed using a scalpel and number 15 blade, a podiatry drill and a spherical podiatry burr
  Interventions: Procedure: Debridement
- Debridement with needle insertion (Sham Comparator): A debridement was followed by the insertion of a 27-gauge needle on a 3 mL syringe that was inserted at 10 to 15 degrees with the bevel facing up approaching from the IPK's right side. The syringe was removed and the IPK was bandaged with a sterile gauze and medical tape.
  Interventions: Procedure: Debridement; Procedure: Needle insertion
- Debridement with physiological water injection (Placebo Comparator): A debridement was followed by the insertion of a 27-gauge needle on a 3 mL syringe that was inserted at 10 to 15 degrees with the bevel facing up approaching from the IPK's right side. The podiatrist pressed completely on the syringe to inject 1 mL of 0.9% sterile sodium chloride water. The syringe was removed and the IPK was bandaged with a sterile gauze and medical tape.
  Interventions: Drug: Physiological water injection; Procedure: Debridement
- Debridement with lidocaine injection (Experimental): A debridement was followed by the insertion of a 27-gauge needle on a 3 mL syringe that was inserted at 10 to 15 degrees with the bevel facing up approaching from the IPK's right side. The podiatrist pressed completely on the syringe to inject 1 mL of 2% lidocaine solution. The syringe was removed and the IPK was bandaged with a sterile gauze and medical tape.
  Interventions: Drug: Lidocaine injection; Procedure: Debridement

INTERVENTIONS:
Drug: Lidocaine injection — 2% (20mg/ml) lidocaine solution
  Arms: Debridement with lidocaine injection
Drug: Physiological water injection — 0.9% sterile sodium chloride water
  Arms: Debridement with physiological water injection
Procedure: Debridement — A debridement was completed using a scalpel and number 15 blade, a podiatry drill and a spherical podiatry burr.
Procedure: Needle insertion — A 27-gauge needle on a 3 mL syringe was inserted at 10 to 15 degrees with the bevel facing up approaching from the IPK's right side
  Arms: Debridement with needle insertion

SUMMARY:
An intractable plantar keratoma (IPK) is a conical thickening of the epidermis' stratum corneum and a common cause of foot pain which can have a significant, detrimental impact on the mobility, quality of life and independence of individuals. Conservative treatments are currently offered to patients with IPK, but they are unsatisfactory since they do not offer a sufficient or permanent reduction of symptoms. The purpose of this study was the evaluation of the feasibility, safety and effectiveness of innovative treatments for intractable plantar keratoma (IPK)

ELIGIBILITY:
Inclusion Criteria:

• Having a painful IPK for at least 3 months

Exclusion Criteria:

* Ongoing pregnancy or breastfeeding
* Severe cardiovascular or neurological disease
* Immunosuppressed status
* Presence of a plantar ulcer
* Allergy to lidocaine
* History of keloid or hypertrophic scar
* Simultaneous painful plantar syndrome unrelated to the presence of an IPK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-07 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain (visual analogue scale) | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 12 months
  Patients were asked to rate their pain level during the seven previous days on the visual analogue scale (VAS). The VAS is a 10 centimeters line anchored at the beginning by "no pain" and at the end by "worst pain imaginable"
Change from baseline in Foot-Function-Index-Revised (FFI-R) | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 12 months
  The Foot Function Index (FFI) measure the impact of foot pathology on function in terms of pain, disability and activity restriction

SECONDARY OUTCOMES:
Change from baseline in size of Intractable plantar keratoma | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 12 months
  IPK's length and width was measured with a millimeter scale ruler used in wound care (accuracy ± 0.1 mm). The depth was estimated with a cotton tip applicator technique measured with the same ruler

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cantin, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Clinique podiatrique de l'Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercier MP, Blanchette V, Cantin V, Brousseau-Foley M. Effectiveness of saline water and lidocaine injection treatment of intractable plantar keratoma: a randomised feasibility study. J Foot Ankle Res. 2021 Apr 13;14(1):30. doi: 10.1186/s13047-021-00467-7. PMID 33849632